CLINICAL TRIAL: NCT03494153
Title: Early Echographic Asystole as a Predictive Factor of Absence of Spontaneous Circulatory Activity Recovery (SCAR) in Prehospital Cardio Respiratory Arrests (CRA) - ACE Study
Brief Title: Early Echographic Asystole as a Predictive Factor of Absence of Spontaneous Circulatory Activity Recovery (SCAR) in Prehospital Cardio Respiratory Arrests (CRA)
Acronym: ACE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0464
Record Dates: First submitted 2018-03-29; First posted 2018-04-11 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Prehospital Cardio-Respiratory Arrests; Spontaneous Circulatory Activity Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non applicable - Non interventional study — Non interventional study

SUMMARY:
Assessment of prognostic performances of CCU in CRA Recovery (CRAR) has already been explored but 1) Only in intra-hospital medicine, 2) in very variable timings. ACE Research focuses on the extra-hospital window and predictive value of Early CCU (within 12 minutes of rescucitation initiation) with ambitious endpoints : curable etiologies identification, early anticipation of ECMO procedures, early anticipation of organ donation process, and evaluation of intrinsic contribution criterion to resuscitation interruption.

The primary objective of ACE study is to investigate the positive predictive value (PPV) of early ultrasound asystole on the absence of CRAR. The secondary objectives are multiple and innovative despite an observational design: impact on the morbi-mortality of the target population (frequency of curable etiologies, pre-therapeutic and therapeutic delays, morbidity...), delay of ECMO implementation of an ECMO (Extracorporeal Membrane Oxygenation), failure rate of organ donation due to overdelays, construction of a multifactorial score associated with CRAR.

DETAILED DESCRIPTION:
Prehospital Cardio-Respiratory Arrests (CRA) represent a significant cause of mortality in France (between 30,000 and 50,000 cases per year) [1]. The prognosis is particularly pejorative, since only 5 to 6% of patients will leave the hospital alive with satisfying neurological condition [2,3]. Their management in France is part of a very singular Primary Care System, based on the medicalization of medical regulation (SAMU) and effectiveness (SMUR) and is based mainly on European recommendations (cardiac massage, ventilation and cardiac rhythm analysis) [4]). European 2015 recommendations advocate for the use of Cardiac Clinical Ultrasound (CCU) in Emergency Medicine, particularly to identify curable causes of CRA. Indeed, CCU is likely to reveal various curable etiologies as tamponade, massive pulmonary embolism, deep hypovolemia or suffocating pneumothorax[5]. Their identification allows the clinician to better adjust his therapeutic strategy and consequently improve patient prognosis.

But its predictive value on the absence of Spontaneous Circulatory Activity Recovery (SCAR) focus clinicians' interest due to its impact on extracorporeal circulation procedures, organ donation or resuscitation interruption guideline. Several studies support the predictive value associated with the absence of mechanical cardiac activity and resuscitation failure [5-10]. However, proof level remains very shaky and transposition to prehospital medicine is clearly impossible (delays, management and environment differ largely). As a corollary, the European Resuscitation Council (ERC) ruled in 2015 that the prognostic performances of ultrasound asystole had not been sufficiently finely measured to consider it as a rigorous criterion for resuscitation interruption, appealing for pivotal studies [4].

ACE French National Trial fits precisely into this bibliographic gap. Our objectives are multiple: assess prognostic value of Early CCU (ECCU; ie. <M12), alone or combined with other clinical parameters (composite prognostic tool combining myocardial and/or electrical activity, capnography, No/Low Flow duration, and clinical profile -sex, age-) on the absence of SCAR ; describe frequency and typology of curable etiologies in the context of CRA, and estimate the possible prognostic impact of early CCU on morbidity and mortality; finally, in case of validation of its prognostic performances, estimate theoretical time savings on ECMO (Extracorporeal Membrane Oxygenation) and organ donation processes.

Multicentric, based on rigorous methodology, high proof-level design and large sample (N=624), ACE wants to be resolutely pragmatic, by associating peripheric hospital and university hospital (Expertise), urban or rural environment (delays and intervention conditions), in order to answer definitely clinicians questioning of the emergency physicians. Continuing in the same vein, we aim a future validation study of a decision-making algorithm for pre-hospital management of CRAs to reduce morbidity and (Randomized Cluster Study in Stepped-Wedge integrating a medico-economic component).

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18yo) presenting extra-hospital CRA.

Exclusion Criteria:

* Resuscitation refusal.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving resuscitation by the SMUR team in an CRA are eligible
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Assess prognostic value of early echographic (ECCU) asystole (i.e. within the first 12 minutes of resuscitation) on resuscitation failure (absence of CRAR). | 1 month
  Patient in CRAR with extra-hospital care

SECONDARY OUTCOMES:
Assess prognostic value of an early echographic (ECCU) asystole (i.e. within the first 12 minutes of resuscitation) on morbi-mortality evaluated at 30 days | 1 month
  Positive predictive value of ultrasound asystole within 12 minutes of the start of specialized CPR on the occurrence of death and/or sequelae at 30 days
Measure variations of the prognostic performances of the extra-hospital ECCU according to their timing of realization, on the absence of CRAR | 1 month
  Sensitive, specificity, negative predictive value, likelihood ratios of early ultrasound asystole to absence of CRAR
Study the link between ultrasound diagnosis and electrocardiogram electrical plots. | 1 month
  Recorded electrical activity patterns:
Creation of a multifactorial composite prognostic score associated with the absence of CRAR | 1 month
  composite score

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pes, Dr, Study Director — Nantes University Hospital
Locations (7):
- France (7):
  - Chu Angers, Angers
  - Chru Brest, Brest
  - Ch Chateaubriant, Châteaubriant
  - Chd Vendee, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - CH Saint-Nazaire, Saint-Nazaire
  - Chru Tours, Tours

REFERENCES:
- [Derived] Papin M, Markarian T, Le Bastard Q, Volteau C, Pes P, Le Conte P, Javaudin F. Inter-rater reliability of point-of-care ultrasound during out-of-hospital cardiac arrest: an ancillary analysis of the observational prospective ACE trial. Resusc Plus. 2025 Dec 13;27:101191. doi: 10.1016/j.resplu.2025.101191. eCollection 2026 Jan. PMID 41583929
- [Derived] Javaudin F, Papin M, Le Bastard Q, Thibault M, Boishardy T, Brau F, Laribi S, Petrovic T, Peluchon T, Markarian T, Volteau C, Arnaudet I, Pes P, Le Conte P. Early point-of-care echocardiography as a predictive factor for absence of return of spontaneous circulatory in out-of-hospital cardiac arrests: A multicentre observational study. Resuscitation. 2024 Oct;203:110373. doi: 10.1016/j.resuscitation.2024.110373. Epub 2024 Aug 21. PMID 39174002
- [Derived] Javaudin F, Pes P, Montassier E, Legrand A, Ordureau A, Volteau C, Arnaudet I, Le Conte P. Early point-of-care focused echocardiographic asystole as a predictive factor for absence of return of spontaneous circulatory in out-of-hospital cardiac arrests: a study protocol for a prospective, multicentre observational study. BMJ Open. 2019 Aug 30;9(8):e027448. doi: 10.1136/bmjopen-2018-027448. PMID 31471433